CLINICAL TRIAL: NCT02642445
Title: Efficacy and Safety of Renal Sympathetic Denervation From The Adventitia on Hypertension in Patients With Primary Aldosteronism
Brief Title: Renal Sympathetic Denervation From The Adventitia on Hypertension
Acronym: RSDAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Principal Investigator, Chuanyu Gao, Principal Investigator, Henan Institute of Cardiovascular Epidemiology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HenanICE201502
Record Dates: First submitted 2015-12-19; First posted 2015-12-30 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Primary Aldosteronism Due to Aldosterone Producing Adenoma
Keywords: Renal sympathetic denervation;hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Renal Sympathetic Denervation (Experimental): Renal sympathetic Denervation are conducted from the adventitia of renal artery
  Interventions: Device: Renal Sympathetic Denervation
- Control Group (No Intervention): Renal Sympathetic Denervation are not conducted in control group.

INTERVENTIONS:
Device: Renal Sympathetic Denervation — We applied a ablation catheter for discrete radiofrequency ablations of 8 W or less and lasting up to 2 min each to obtain up to four-six ablations separated both longitudinally and rotationally from the adventitia
  Arms: Renal Sympathetic Denervation

SUMMARY:
Renal sympathetic denervation from the intima of renal arteries has become an important method for the treatment of resistant hypertension, but renal sympathetic nerve are mainly located in the adventitia, and there is no report about renal sympathetic denervation from the renal adventitia. Primary aldosteronism is an important factor of secondary hypertension, tumor aldosterone in unilateral adrenal can increase the concentration of plasma aldosterone, in some patients blood pressure control is still not desirable after resection of tumor aldosterone. This study intends to conduct renal sympathetic denervation ablation from the adventitia to observe its efficacy and safety on blood pressure of patients with primary aldosterone.

DETAILED DESCRIPTION:
Renal sympathetic denervation from the intima of renal arteries has become an important method for the treatment of resistant hypertension, but renal sympathetic nerve are mainly located in the adventitia, and there is no report about renal sympathetic denervation from the renal adventitia. Primary aldosteronism is an important factor of secondary hypertension, tumor aldosterone in unilateral adrenal can increase the concentration of plasma aldosterone, in some patients blood pressure control is still not desirable after resection of tumor aldosterone.

This study intends to conduct renal sympathetic denervation ablation（RDN）from the adventitia to observe its efficacy and safety on blood pressure of patients with primary aldosterone.

ELIGIBILITY:
Inclusion Criteria:

1. . Renal artery diameter ≥4 mm and Length ≥20 mm;
2. . 18 years old ≤ age ≤ 70 years old;
3. . Specific diagnosis of adrenal adenoma and primary aldosteronism before the patients are enrolled in the study;
4. . Clinic systolic blood pressure≥160 mmHg and/or diastolic blood pressure≥100 mmHg (patients with type 2 diabetes: clinic systolic blood pressure≥150 mmHg and/or diastolic blood pressure≥95 mmHg) .
5. . 24 hours ambulatory blood pressure (SBP/DBP)≥140 and/or 90 mmHg;
6. . Estimated GFR (eGFR)≥45 ml/min / 1.73 m2.

Exclusion Criteria:

1. . Renal artery abnormalities include: either side renal arterial blood flow mechanics or anatomical obvious stenosis (≥50% ); Underwent renal artery balloon angioplasty or inserting a stent; Renal artery anatomy apparently is unusual to insert catheter;
2. . Cardiovascular instability includes: myocardial infarction in six months, unstable angina or cerebrovascular disease; Thrombus or unstable plaques in the arteries with extensive atherosclerosis; Hemodynamic apparently change in patients with heart valve disease;
3. . The patients with typeⅠdiabetes;
4. . Other serious organic disease;
5. . Participated in other clinical research.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-12; Primary Completion 2019-03-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Systolic Blood Pressure at 6 months,12 months, 18 months | at 6 months,12 months,18 months
  The Change of Systolic Blood Pressure from Baseline to 6 months,12 months, 18 months

SECONDARY OUTCOMES:
Change from Baseline Renin at 6 months,12 months, 18 months | at 6 months,12 months,18 months
  The Change of Renin from Baseline to 6 months,12 months, 18 months
Change from Baseline aldosterone at 6 months,12 months, 18 months | at 6 months,12 months,18 months
  The Change of aldosterone from Baseline to 6 months,12 months, 18 months

CONTACTS AND LOCATIONS:
Overall Officials: ChuanYu Gao, Dr., Principal Investigator — Henan Institute of Cardiovascular Epidemiology; Dayi Hu, Dr., Principal Investigator — Henan Institute of Cardiovascular Epidemiology
Locations (1):
- Zhengzhou university People's Hospital, Zhengzhou, Henan, China